CLINICAL TRIAL: NCT06598410
Title: The Effect of Playing Digital Games and Watching Cartoons on Children&Amp;#39;s Pain, Fear, and Anxiety Levels During Suturing in Pediatric Emergency Unit
Brief Title: Playing Digital Games and Watching Cartoons on Children&Amp;#39;s Pain, Fear, and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Atiye Karakul, Assoc. Prof., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/76
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pain; Fear; Anxiety; Children; Emergency
Keywords: pain; fear; anxiety; emergency; pediatri
MeSH Terms: conditions — Pain; Anxiety Disorders; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digital Gaming (Experimental): Children will play digital games during suturing in the Paediatric Emergency Unit
  Interventions: Other: Digital gaming
- Watching Cartoon (Experimental): Children will watching cartoon during suturing in the Paediatric Emergency Unit
  Interventions: Other: watching cartoon
- Control (No Intervention): Children will not be subjected to any form of distraction

INTERVENTIONS:
Other: Digital gaming — Children in this group will be allowed to play digital games 5 minutes before the procedure starts. They will continue to play the game during the procedure.
  Arms: Digital Gaming
Other: watching cartoon — Children in this group will be shown a cartoon film 5 minutes before the procedure. They will continue to play the game during the procedure.
  Arms: Watching Cartoon

SUMMARY:
The study was planned as a randomized controlled experimental study to determine the effect of playing digital games and watching cartoons on the pain, fear, and anxiety levels of children during suturing in the pediatric emergency unit. The population of the study, which is planned as a randomized controlled experimental study, will consist of children between the ages of 5-10 who apply to the Trauma Unit of the Pediatric Emergency Unit of Tarsus State Hospital and undergo suturing.

As a result of the Power analysis (G*Power 3.1.9.2); effect size = 1.136, 95% confidence interval, 95% power, it was calculated that a total of 66 children, at least 22 in each group, should be included. Considering that there may be dropout and confounding variables in the research process, it was determined as 90 children in total, with 30 children in each group.

Implementation Stage 1: A pool of cartoons that can be watched and digital games that can be played, suitable for the level of the child in the 5-10 age group, will be created by the researchers by taking the opinion of the relevant experts. The created children's cartoon and digital game pool will be sent to experts in the field (child development specialist, child psychiatrist, child nurse).

Stage 2: A pilot study will be conducted with 10 children to evaluate the suitability of data collection forms, digital games and cartoons for children.

Stage 3: The children and family members in the sample group will be informed about how the application will be carried out and about the research, and written permission will be obtained from the family and verbal permission will be obtained from the child.

It will be ensured that the children in all groups will have their parents with them during the procedure.

Stage 4: Children who meet the sample selection criteria will be divided into 3 groups (1st study group, 2nd study group, and 3rd group control group) through a computerized programme.

Stage 5: The data collection form in the research will be applied to the children in the sample group before the procedure.

6th Stage: The pain, fear and anxiety of the children in all groups before the procedure will be evaluated by the child, parent and nurse.

DETAILED DESCRIPTION:
Children experience a traumatic process if cuts occur anywhere on their body after an accident. It has been reported that nursing interventions applied during incision suturing relieve the anxiety and fears of the child. Two main ways are defined as pharmacological and non-pharmacological methods in pain and anxiety management. Therefore, standards have not yet been established for their inclusion in daily patient care. Non-pharmacological methods aim to reduce fear, anxiety, and pain and to give children a sense of control. Both physical and cognitive behavioral approaches are necessary to provide a comfortable environment for children. It is also important to use non-pharmacological interventions during medical procedures to reduce the stress experienced by parents. Nurses can apply these methods independently and encourage family members to participate in patient care actively. Visual distractions minimize pain and also allow action to be taken in an emergency. Various games and cartoons allow the child to express their fears, misconceptions, and anxieties in their own way, both verbally and non-verbally, thus helping the child to cope with stressful situations.

The study was planned as a randomized controlled experimental study to determine the effect of playing digital games and watching cartoons on the pain, fear, and anxiety levels of children during suturing in the pediatric emergency unit. The population of the study, which is planned as a randomized controlled experimental study, will consist of children between the ages of 5-10 who apply to the Trauma Unit of the Pediatric Emergency Unit of Tarsus State Hospital and undergo suturing.

While determining the sample size of the study, as the result of the literature review to determine the effect size sample size, Kavlakcı (2020) 'The Effect of Digital Game Playing on Pain, Fear and Anxiety Levels During Suturing in Children: A Randomised Controlled Study' was taken as a basis. As a result of the Power analysis (G*Power 3.1.9.2); effect size = 1.136, 95% confidence interval, 95% power, it was calculated that a total of 66 children, at least 22 in each group, should be included. Considering that there may be dropout and confounding variables in the research process, it was determined as 90 children in total, with 30 children in each group.

The data of the research will be collected using the following data collection tool:

Introductory Information Form: It consists of a total of 15 questions, including sociodemographic characteristics (13) questions and (2) questions about the procedure, prepared in line with the literature.

2. Child Fear Scale: The scale was developed by Thurillet et al. to evaluate the fears of children based on the self-report of children aged 4-12 years. Turkish validity and reliability study was conducted by Tavşan et al. The scale consists of six facial expressions. The scale grades fear with a score ranging from 0 to 10 (gradually graded two by two) consistent with pain rating scales. The first facial expression indicates that there is no fear, the fear increases as you go from right to left, and the sixth facial expression indicates that the level of fear is the highest. A statistically significant positive and very high correlation was obtained between the Fear Scale and the Child Fear Scale. The high correlation value between the two forms shows that the child form is valid. The content validity index and item-coverage validity index values of the scale were found to be 0.98. A very good statistically significant agreement was achieved between the Fear Scale and the Child Fear Scale. Permission for the use of the scale was obtained from the author via e-mail.

3. Child Anxiety Scale-Dispositional Scale (CAS-D) :The Turkish validity and reliability study of the Child Anxiety Scale-Dispositional (CAS-D) scale developed by Ersig et al. to measure the anxiety levels of children aged 4-10 years was conducted by Gerçeker et al. The CAS-D scale is shaped like a thermometer with a light bulb at the bottom and horizontal lines with intervals going upwards. In this scale for children aged 4-10 years, children are asked 'Imagine that all your anxious or nervous feelings are at the bulb or bottom of the thermometer' or 'If you are a little anxious or nervous, the feelings may go up a little on the thermometer. If you are very, very anxious, or nervous, emotions can go all the way to the top. Put a line on the thermometer showing how anxious or nervous you are. In order to measure state anxiety (CAS-D), the child is asked to tick how he/she feels 'right now'. The score can vary between 0-10. Permission for the use of the scale was obtained from the author via e-mail.

4. Wong-Baker Pain Scale: It was developed by Donna Wong and Connie Morain Baker in 1980 and adapted again in 1983 to measure the pain levels of pediatric patients. There are 6 facial expressions scored between 0-5. In the Wong-Baker Scale, there are facial expressions indicating the increasing degree of pain from 0 to 5 from left to right.

5. Life Findings Follow-up Form: It was prepared to record the heart rate, saturation value and respiration values of the children when they came to the trauma unit before the procedure and the vital signs measured immediately after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Between 5-10 years old
* Suture removal will be applied
* Number of sutures 3 or more
* volunteering to participate in the study.

Exclusion Criteria:

* No previous suturing procedure
* Suturing to be applied to the hand, arm area
* The child has visual, hearing and intellectual disabilities
* Having a physical problem that prevents them from playing digital games

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
pain level | 1 hour
  Wong Baker Pain Scale: It was developed by Donna Wong and Connie Morain Baker in 1980 and adapted again in 1983 to measure the pain levels of paediatric patients. There are 6 facial expressions scored between 0-5. In the Wong-Baker Scale, there are facial expressions indicating the degree of pain increasing from 0 to 5 from left to right.
fear | 1 hour
  Child Fear Scale: The scale was developed by Thurillet et al. It was developed to evaluate children's fears based on self-report of children aged 4-12 years. The scale consists of six facial expressions. The scale grades fear with a score ranging from 0 to 10 (gradually graded two by two) consistent with pain rating scales. The first facial expression shows that there is no fear, the fear increases as you go from right to left, and the sixth facial expression shows that the level of fear is the highest. A statistically significant positive and very high correlation was obtained between the Fear Scale and the Child Fear Scale (r=0.973; p;0.001). The high correlation value between the two forms shows that the child form is valid.
anxiety | 1 hour
  Child Anxiety Scale-Dispositional Scale (CAS-D): It was developed by Ersig et al. (2013) to measure the anxiety levels of children aged 4-10 years. The CAS-D scale is shaped like a thermometer with a light bulb at the bottom and horizontal lines with intervals going upwards. In this scale for children aged 4-10 years, children are asked 'Imagine that all your anxious or nervous feelings are at the bulb or bottom of the thermometer' or 'If you are a little worried or nervous, the feelings may go up a little on the thermometer. If you are very, very anxious or nervous, emotions can go all the way to the top. Put a line on the thermometer showing how anxious or nervous you are'. In order to measure state anxiety (CAS-D), the child is asked to tick how he/she feels 'right now'. The score can range from 0-10.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Tarsus University, Mersin
  - Tarsus University, Tarsus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Duzkaya DS, Bozkurt G, Ulupinar S, Uysal G, Ucar S, Uysalol M. The Effect of a Cartoon and an Information Video About Intravenous Insertion on Pain and Fear in Children Aged 6 to 12 Years in the Pediatric Emergency Unit: A Randomized Controlled Trial. J Emerg Nurs. 2021 Jan;47(1):76-87. doi: 10.1016/j.jen.2020.04.011. Epub 2020 Jul 18. PMID 32690314
- [Result] Topan, A., Bayram, D. ve Ayyıldız, T. K. (2019) Pediatrik Acil Servise Başvuran 0- 18 Yaş Grubu Olgular: Retrospektif İnceleme. İzmir Kâtip Çelebi Üniversitesi Sağlık Bilimleri Fakültesi Dergisi. Vol. 4(3-1), ss. 300-305.
- [Result] Yıldız S. Acile başvuran çocuk ve aileye psikososyal yaklaşım. Atatürk Üniversitesi Hemşirelik Yüksekokulu Dergisi. 2006; 9(3); 69-76
- [Result] Thurillet S, Bahans C, Wood C, Bougnard S, Labrunie A, Messager V, Toniolo J, Beloni P, Fourcade L. Psychometric properties of a self-assessment fear scale in children aged 4 to 12 years. Scary Scale. J Pediatr Nurs. 2022 Jul-Aug;65:108-115. doi: 10.1016/j.pedn.2022.02.020. Epub 2022 Mar 14. PMID 35300885
- [Result] HasasnTehrani, T., Pakzad, A., Mohammadi, F., Tapak, L., &Azmamoun, H. (2022). Effect of Pre-endoscopyPreparation Program on Children'sAnxietyandParentalSatisfaction: A Clinical Trial Study. EvidenceBasedCare, 11(4), 48-54.
- [Result] Guerrero-Marquez G, Martinez-Serrano A, Miguez-Navarro C, Lopez-Miron JA, Espartosa-Larrayad M. [Knowledge of nurses about medication doses at pediatric urgency departament]. Enferm Clin. 2016 Jul-Aug;26(4):213-9. doi: 10.1016/j.enfcli.2016.04.009. Epub 2016 Jun 11. Spanish. PMID 27297176
- [Result] Chen YJ, Cheng SF, Lee PC, Lai CH, Hou IC, Chen CW. Distraction using virtual reality for children during intravenous injections in an emergency department: A randomised trial. J Clin Nurs. 2020 Feb;29(3-4):503-510. doi: 10.1111/jocn.15088. Epub 2019 Dec 4. PMID 31715039
- [Result] Capua T, Kama ZB, Rimon A. The influence of an accredited pediatric emergency medicine program on the management of pediatric pain and anxiety. Isr J Health Policy Res. 2018 Mar 21;7(1):17. doi: 10.1186/s13584-018-0211-6. PMID 29562929
- [Result] Abuqamar M, Arabiat DH, Holmes S. Parents' Perceived Satisfaction of Care, Communication and Environment of the Pediatric Intensive Care Units at a Tertiary Children's Hospital. J Pediatr Nurs. 2016 May-Jun;31(3):e177-84. doi: 10.1016/j.pedn.2015.12.009. Epub 2016 Jan 20. PMID 26803562